CLINICAL TRIAL: NCT06875323
Title: CASA and FostrSpace: Systems Delivery of Digital Substance Use Prevention Tools to Foster Youth
Brief Title: FostrSpace-CASA R61/R33
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R61DA059860-01 (NIH); R61DA059860 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Substance Use
Keywords: Foster youth; Substance use; mHealth
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InfoECHO (Experimental): CASA volunteers will attend a six 90-minute/biweekly co-occurring SU and trauma ECHO trainings.
  Interventions: Other: ECHO-FostrSpace
- InfoOnly (Other): CASA volunteers will attend a one-time 30-60 minute co-occurring SU and trauma ECHO training.
  Interventions: Other: Informational Session

INTERVENTIONS:
Other: ECHO-FostrSpace — Six ECHO-FostrSpace session training for CASA volunteers.
  Arms: InfoECHO
Other: Informational Session — One ECHO-FostrSpace session training for CASA volunteers.
  Arms: InfoOnly

SUMMARY:
The purpose of this study is to understand how an online digital health application (app) called FostrSpace can reduce substance use among youth (ages 13-20 years old) in foster care.

DETAILED DESCRIPTION:
The goal of this clinical trial is to identify gaps in substance use prevention across existing CASA trainings and the FostrSpace app for foster youth and test how substance use trainings for CASA volunteers could help facilitate FostrSace app referrals to reduce and prevent substance use among CASA youth.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults will be eligible if they are age 13-20, are proficient in English, have an assigned CASA worker, and have a device with web access.
* CASAs (ages 18 and over) will be eligible if they are assigned to a youth between the ages of 13- 20.

Exclusion Criteria:

* Youth: Exclusion criteria include being non-English speaking, being within 3 months of ending with CASA services, cognitive impairment that precludes ability to provide informed consent.
* CASA: Exclusion criteria include being non-English speaking and working with a youth who is within 3 months of ending with CASA services.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Drug Use | baseline
  The Texas Christian University (TCU) drug screen with opioid supplement is used to gather detailed information about drug and opioid use.
Rate of Cigarette Use | baseline
  The Cigarette smoking and vaping/e-cigarette use is used to gather detailed information about nicotine and/or cannabis use.

SECONDARY OUTCOMES:
The Alcohol and Marijuana Expectancy Questionnaire | baseline
  The Alcohol and Marijuana Expectancy questionnaire is used to measure positive and negative expectancies about affective, cognitive and behavioral effects of alcohol and cannabis use. Items are rated from 1-5 scale and higher scores indicate negative alcohol and marijuana expectancies.
The Brief Young Adult Alcohol Consequences Questionnaire | baseline
  The Brief Young Adult Alcohol Consequences Questionnaire is used to assess the severity of alcohol consumption. Higher scores indicate greater severity of consequences associated with alcohol consumption.
The Brief Marijuana Consequences Questionnaire | baseline
  The Brief Marijuana Consequences Questionnaire is used to assess the severity of marijuana consumption. Higher scores indicate greater severity of consequences associated with marijuana consumption.
The Brief Symptom Inventory | baseline
  Brief Symptom Inventory is used to measure depression, anxiety and somatization symptoms to assess for psychiatry distress. Index ranging from 0 to 72 with cut-score of 11 as indication of psychiatric distress.

OTHER OUTCOMES:
CASA Background Characteristics | baseline
  Demographics questionnaire used to gather standard demographics (e.g., age, gender, race) and information such as state agency involvement (e.g., age at first contact with child welfare, number of out-of-home placements, length of time worked with a CASA), immigration status.
Arrest and Treatment | baseline
  The Arrest and treatment history (ATH) questionnaire is used to gather information about past juvenile legal system contact (arrest, probation, detention), mental health (MH) and substance use (SU) diagnoses, and past services utilization for SU and/or MH (inpatient, residential, outpatient).
Youth Background Characteristics | baseline
  Youth's living situation questionnaire will be used to gather information related to the youth's living situation over the past 4 months (e.g., in the community, residential treatment, or other living situation).
Social Determinants of Health | baseline
  We will administer an 18-item yes/no questionnaire to gather information on what youth perceive as most relevant and important social determinants of health items for foster youth (i.e., employment, food, family, healthcare, housing, legal, education, safety at school/work, transportation, "other" needs).
Therapeutic Alliance | baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with provider) over time. Scores range from 12-84 with higher scores indicating greater perceived therapeutic alliance.
Youth/CASA Relationship | baseline
  Frequency and quality of CASA-youth conversations about substance use: For frequency, we will adapt an item from a validated measure of parent-child communication about sex used in previous studies45 "How many times have you and your CASA talked about [alcohol, marijuana, cocaine]" (each drug asked separately). For quality, we will use one-item from the scale that assesses perceived helpfulness 'How helpful do you think your discussions about alcohol and/or drugs were?' and one-item that assesses perceived comfort 'How comfortable are you with these discussions about alcohol and/or drugs with your [CASA youth] or [CASA].
Trauma | baseline
  6: deidentified assessment of Adverse Childhood Experiences (10 items) and Related Life Events (7 items).
Ethnic Identity | baseline
  The Scale of Ethnic Experience is used to measures youth ethnicity-related cognitive constructs (e.g., perceptions of their own ethnic group, ethnic group belonging) in four domains: Ethnic Identity(12-items; α =.87); Perceived Discrimination (9-items; α = .91); Mainstream Comfort (6-items; α=.87); and Social Affiliation (5-items; α =.83). Items rated on a scale from 1 (strongly disagree) to 5(strongly agree).
Stigma | baseline
  The Social Distance Scale (SDS) is used to assess a person's willingness to interact with others with mental illness (SDS) or substance users (SDS-SU).
Peer Substance Use | baseline
  The Monitoring the Future is used to assess how many close friends are using alcohol, cannabis and other drugs occasionally and regularly.
Background Characteristics | baseline
  A Demographics Questionnaire is used to gather standard demographics (e.g., age, gender, race) and information about employment, number of years as CASA volunteer, length of time known current foster youth, immigration status, country of origin.
Substance use prevention related knowledge, beliefs, attitudes and self efficacy | baseline
  Beliefs about youth SU will be measured using an adapted 9 item perceived risk of SU measure used in studies of similar risk perceptions (among parents) associated with youth substance use. Items such as "If your youth were to use alcohol more than once a week, what do you think are the chances of them becoming (for example) addicted to alcohol, developing cancer (or lung cancer for drugs that can be smoked), experiencing brain injury etc.
Compassion Satisfaction and Fatigue | 30 days post baseline, 60 days post baseline
  The Professional Quality of Life will be used to gather information about compassion satisfaction and compassion fatigue.
FostrSpace App Utilization | baseline, 30 days post baseline, 60 days post baseline
  Number of app log-in's, days of use, time spent using app, number and type of features used e.g.,chat use (peer/FAB), chat use (navigator), number of clicks on SU prevention content (e.g., SU resources requested, peer "adulting 101" SU prevention video watched), requested navigator support (yes/no), requested navigator support about SU (yes/no), requested teletherapy [primary presenting need, type of intervention, e.g., primary SU or MH or co-occurring, modality of intervention (individual, group, family), number and frequency of sessions received].
Psychiatric Symptoms | baseline
  The Emotional Wellness Questionnaire is used to assess psychiatric symptoms (e.g., depression, anxiety, mania) and substance use.
FostrSpace Usability | 30 days post baseline, 60 days post baseline
  The System Usability Scale (SUS) is used to gather information about the overall usability of web applications.
  10- item measure widely used for web applications and proven superior to other measures. SUS yields a single number representing a composite measures of the overall usability of the system being studied60,61. Scores will be compared to established norms for levels of usability. Our goal is a score of 80 (top 10% of scores), which reflects excellent usability, and is associated with recommending the product to a friend.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No